CLINICAL TRIAL: NCT06030622
Title: Phase 2A Pilot Trial of Metformin, Digoxin, Simvastatin (C3) in Combination With Gemcitabine in Subjects With Recurrent / Refractory Metastatic Advanced Pancreatic Cancer
Brief Title: Phase 2A Pilot C3 Trial of Recurrent/Refractory Metastatic Advanced Pancreatic Cancer
Acronym: C3
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Mohan Preet, Oncologist, State University of New York - Downstate Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1727019-4
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer Metastatic
Keywords: C3 trial; metformin; simvastatin; digoxin; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Metformin; Simvastatin; Digoxin; Single Person

STUDY DESIGN:
Intervention Model Description: The treatment plan is as follows: The first 3 patients enrolled in the study, will receive metformin (850 mg twice a day), digoxin (0.25 mg once a day), and simvastatin (20 mg once a day) for 28 days. If no toxic effects, the remaining 22 patients will be enrolled. Patients will be provided C3 medications every 28 days and will continue on the C3 medication for at least 2 years, or until death or recurrence/advancement of the disease. If more than one patient develops a toxic event, the dose will be reduced to metformin 850 mg/day, simvastatin 5 mg/day, and digoxin 0.0625 mg/day. If no further toxicities, then the remaining patients will receive the lower dose. If however, more than two patients develop a toxic event, then study discontinuation will be considered. If patients decline first line therapy (Gemcitabine), they will be offered the choice of C3 medications only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gemcitabine and C3 (Combination Digoxin, Simvastatin, and Metformin) (Experimental): Study participants will be offered metformin (850 mg twice a day), digoxin (0.25 mg once a day), and simvastatin (20 mg once a day) combination (C3) and Gemcitabine.
  Interventions: Drug: Gemcitabine and C3 (Metformin, Simvastatin, and Digoxin)
- C3 (Combination Digoxin, Simvastatin, and Metformin) only (Experimental): Study participants will be offered C3 only metformin (850 mg twice a day), digoxin (0.25 mg once a day), and simvastatin (20 mg once a day) combination (C3) if they decline Gemcitabine.
  Interventions: Drug: C3 (Metformin, Simvastatin, and Digoxin) only

INTERVENTIONS:
Drug: Gemcitabine and C3 (Metformin, Simvastatin, and Digoxin) — Combination treatment of Metformin, Simvastatin and Digoxin with Gemcitabine (Arm 1)
  Other Names: Glucophage, Zocor, Digitalis, Gemzar
  Arms: Gemcitabine and C3 (Combination Digoxin, Simvastatin, and Metformin)
Drug: C3 (Metformin, Simvastatin, and Digoxin) only — C3 only (Metformin, Simvastatin, and Digoxin) if patients decline Gemcitabine (Arm 2).
  Other Names: Glucophage, Zocor, Digitalis
  Arms: C3 (Combination Digoxin, Simvastatin, and Metformin) only

SUMMARY:
The goals of this trial are: 1) To evaluate the safety and tolerability of C3 administration with Gemcitabine; and 2) To assess the disease response following C3 administration with Gemcitabine. The main question it aims to answer are: 1) Is C3 in combination with Gemcitabine safe, tolerable, and effective for reducing improving advanced stage pancreatic cancer? and 2) Can C3 in combination with Gemcitabine prolong the lives of patients with advanced stage pancreatic cancer. Participants will receive a combination of metformin (850 mg twice a day), digoxin (0.25 mg once a day), and simvastatin (20 mg once a day), also known as C3, and Gemcitabine (as per standard of care) for 2 years. If patients decline Gemcitabine, they will be offered the C3 medications only.

DETAILED DESCRIPTION:
Background. Pancreatic Ductal Adenocarcinoma (PDAC) is one of the deadliest cancers and ranks fourth in cancer-related deaths in the United States. It is among the 10 most commonly diagnosed cancers (9th in women and 10th in men), with approximately 56,770 new cases and 45,750 deaths in 2019. Current therapy for advanced disease includes the use of medications such as Gemcitabine, Erlotinib, Capecitabine, or combination treatments such as 5-fluorouracil, irinotecan, and oxaliplatin; or Gemcitabine and nab-paclitaxel. These standard of care medications have a survival advantage of less than six months in patients with advanced metastatic disease. Recent studies have shown that the use of metformin and simvastatin in 15,099 patients with pancreatic cancer significantly improved their survival.

Study Design/Methods. Based on those prior studies, the investigators will conduct an open-label, single-center, phase 2, feasibility trial of a combined metformin, digoxin, and simvastatin (C3) in 25 subjects with recurrent/refractory metastatic pancreatic cancer in order to evaluate their safety and tolerability. Patients who were previously treated for advanced pancreatic disease with no significant improvements in their disease, will be enrolled in this trial. C3 will be given as oral pills as described in recommended package insert safe levels in addition to their standard of care medication, Gemcitabine.

Study Interventions/Treatment Plan. The treatment plan is as follows: The first 3 patients enrolled in the study, will receive metformin (850 mg twice a day), digoxin (0.25 mg once a day), and simvastatin (20 mg once a day) for 28 days. If no toxic effects, the remaining 22 patients will be enrolled. Patients will be provided C3 medications every 28 days and will continue on the C3 medication for at least 2 years, or until death or recurrence/advancement of the disease. If more than one patient develops a toxic event, the dose will be reduced to metformin 850 mg/day, simvastatin 5 mg/day, and digoxin 0.0625 mg/day. If no further toxicities, then the remaining patients will receive the lower dose. If however, more than two patients develop a toxic event, then study discontinuation will be considered. If patients decline first line treatment (Gemcitabine), they will be offered a choice of C3 medications only.

Safety and Disease Response Assessments. During the conduct of the study, safety assessments will be conducted including physical examination, vital signs monitoring, performance status evaluation, blood CBC/serum chemistry, digoxin levels, toxicity assessment, and radiological tumor assessment. Disease response will be assessed using radiologic tumor assessments, and levels of biomarkers.

Objectives and Endpoints. The Primary Objectives are: 1) To evaluate the safety and tolerability of C3 administration with Gemcitabine. Endpoint and Outcome Measures: Adverse events and abnormalities in laboratory test values, markedly abnormal vital sign measurements; and 2) To assess disease response following C3 administration with Gemcitabine. Endpoint and Outcome Measures: Radiologic tumor assessment at baseline and quarterly thereafter. The Secondary Objectives are: 1) To assess levels of tumor biomarkers. Endpoint and Outcome Measures: Biomarker levels will be determined at baseline and at 2 months after C3 treatment; and 2) To assess molecular changes in biomarkers induced by C3 administration. Endpoint and Outcome Measures: Molecular expressions of tumor biomarkers such as BIRC5, CA19-9, and CEA at baseline, and 2 months after C3 treatment.

Given the safety profile of C3 in thousands of patients, the investigators anticipate that it will significantly improve the disease outcomes and prolong the lives of patients with metastatic advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 years with histologically confirmed pancreatic cancer.
2. Refractory, intolerant to, or with disease progression after at least one standard of care regimen.
3. ECOG performance status (PS) 0-1.
4. Pretreatment biopsy and/or adequate archival tissue available for BIRC5 protein level evaluation.
5. Adequate organ and marrow function: absolute granulocyte count ≥1,000/mm3, platelets ≥100,000/mm3, total bilirubin ≤ institutional upper normal limit, AST/ALT ≤2x institutional upper limit of normal, and creatinine <1.5 mg/dL or calculated creatinine clearance > 60ml / min (Cockcroft-Gault Equation).
6. Subject has recovered to CTCAE Grade 1 (except for alopecia) or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade 2 or better.
7. If participant of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry. Serum pregnancy tests will be conducted at the time of screening, when other blood draws are obtained (See Appendix III: Time-Table of Procedures).
8. Ability to understand and the willingness to sign a written informed protocol specific consent.
9. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. No known active infections at the time of enrollment as determined by negative procalcitonin level.

Exclusion Criteria:

1. Anti-cancer chemotherapy, biologic therapy or immunotherapy within 3 weeks or radiation therapy within 2 weeks of first investigational product administration.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
3. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
4. Known history of rhabdomyolysis.
5. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the Investigator.
6. Known chronic Hepatitis B or C infection.
7. Have current active infection requiring systemic antibiotic treatment.
8. History of severe allergic, anaphylactic, hypersensitivity reactions or previous intolerance to Metformin, Simvastatin, and/or Digoxin.
9. Patients with significant cardiac disease or condition listed below (unless clearance obtained by cardiology):

   1. Wolff-Parkinson-White Syndrome.
   2. Previous MI within last 6 months of C1D1.
   3. Evidence of residual electrographic pattern consistent with heart block., for example atrio-ventricular (AV) heart block (currently ongoing).
   4. History of ventricular fibrillation.
   5. Sick Sinus Syndrome or Sinus bradycardia thought to be caused by sinus node disease, unless effectively treated.
   6. Heart failure with preserved LVEF, including constructive pericarditis, and amyloid heart disease.
10. Acute cor pulmonale, restrictive cardiomyopathy, and Amyloid heart muscle disease.
11. Participants of childbearing potential who are found to be pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) or nursing.
12. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or trial results.
13. Cognitively impaired and diminished capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-17 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Safety and tolerability | 28 days
  Number of participants with treatment-related Adverse Events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Secondary Outcome: Biomarkers | Before and 2 months after C3 treatment
  Tumor biomarkers as assessed by levels of BIRC5, CA19-9, CEA.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Preet, MD, Principal Investigator — SUNY Downstate Health Sciences University
Locations (1):
- SUNY Downstate Health Sciences University, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared will include: patient demographics, vital signs, medical history, clinical laboratory tests, examination results, non-medication treatments (surgeries, procedures), physical examinations, and any adverse events related or unrelated to the investigational product, maximum tolerable dose (MTD), dose-limiting toxicities (DLT), all diagnoses, etc. All secondary outcomes (biomarkers, tumor size). All sensitive information will be secured using compliant encryption software and adequate physical security and operational controls. To de-identify the data, codes that participants will be removed from the data set and birth date will be converted to age to avoid "deductive disclosure" of participants. The Principal Investigator will make the final, de-identified, study data set and associated documentation available to the statistician. The study team will develop a data sharing agreement that provides for a commitment to using the data only for research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: September 30, 2024 to September 30, 2026
Access Criteria: Data will be made available to the general public only through presentations and publications with no identifiers. Data will be shared in continuing education programs at a national and international level. Data will be shared in appropriate forums. All Protected Health Information (PHI) will be restricted to the PI and their research designees. Researchers who seek to obtain data will submit a request to the PI and IRB for approval. However, no PHI will be shared. The PI will ensure that shared data are protected. Data to be transferred for additional analyses will be de-identified and an agreement for confidentiality of data will be obtained from the secondary user who must agree to protect the data. This will include communicating the data protection plan; determining whether the original consent agreement limited the use of the data in future studies; and obtaining a written and binding agreement from the recipient that the data are bound by all of the agreed conditions.
URL: https://www.downstate.edu